CLINICAL TRIAL: NCT02629874
Title: Randomized Double Blind Placebo-controlled Clinical Safety, Tolerability and Pharmacokinetic/-Dynamic Study on the Effects of Escalating Single Intravenous Doses of EA-230 on the Innate Immune Response During Experimental Human Endotoxemia
Brief Title: PK/PD of EA-230 During Endotoxemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Exponential Biotherapies Inc. (Industry)
Responsible Party: Principal Investigator, Peter Pickkers, prof. dr., Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: EBI-EA230-LPS-2014
Record Dates: First submitted 2015-11-16; First posted 2015-12-14 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Endotoxemia; Systemic Inflammatory Response
Keywords: EA-230; Inflammatory response; Kidney Injury; Endotoxemia
MeSH Terms: conditions — Endotoxemia | interventions — alanyl-glutaminyl-glycyl-valine; Endotoxins; Lipopolysaccharides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- EA-230 (30mg/kg) (Active Comparator): Subjects will receive EA-230, 30 mg/kg
  Interventions: Drug: EA-230; Drug: Endotoxin
- EA-230 (90mg/kg) (Active Comparator): Subjects will receive EA-230, 90 mg/kg
  Interventions: Drug: EA-230; Drug: Endotoxin
- EA-230 (180mg/kg) (Active Comparator): Subjects will receive EA-230, 180 mg/kg
  Interventions: Drug: EA-230; Drug: Endotoxin
- Placebo (Placebo Comparator): subjects receive placebo
  Interventions: Drug: Endotoxin; Drug: Placebo

INTERVENTIONS:
Drug: EA-230 — at t=0 30, 90 or 180 mg/kg EA-230 will be administered intravenously over 2 hours.
  Other Names: AQGV
  Arms: EA-230 (180mg/kg); EA-230 (30mg/kg); EA-230 (90mg/kg)
Drug: Endotoxin — at t=0 2ng/kg purified E.Coli endotoxin is administered intravenously
  Other Names: LPS, lipopolysaccharide
Drug: Placebo
  Arms: Placebo

SUMMARY:
EA-230 is a newly developed synthetic compound with anti-inflammatory properties. Pre-clinical data indicate that EA-230 may be a valuable treatment for systemic inflammation resulting from a variety of causes such as surgery, trauma, infection, irradiation and others. Although previous studies in healthy volunteers have shown an excellent safety profile, the safety and tolerability of higher doses administered per continuous infusion need to be investigated. Also, the dose-effect relation on systemic inflammation needs to be further elucidated before a phase II trial in patients can be commenced.

DETAILED DESCRIPTION:
Although the immune system is essential to survival, a variety of diseases originate from inappropriate activation of the immune response. Besides a range of auto-inflammatory disease like rheumatoid arthritis, inappropriate or undesirable activation of the immune system can occur during infectious diseases like sepsis, after major surgery like cardiac artery bypass grafting, after radiation therapy in the treatment of cancer, or after organ transplantation.

For auto-inflammatory diseases, in the last decades therapies have come available that specifically target parts of the immune system. The development of 'biologicals', recombinant antibodies that specifically block one antigen or receptor, has had an enormous impact on the treatment of chronic autoimmune diseases. However, these treatments have been shown not to be effective in other types of (acute) systemic inflammation, like sepsis.

Of the many downstream consequences of exaggerated inflammatory response, organ injury and failure is the most serious, most often involving the kidneys. This also holds true for cardiac surgery with cardiopulmonary bypass, in which various factors, including the inflammatory cascade, cause a temporarily decline or even permanent loss of renal function. As kidney failure is an independent prognostic factor for mortality in critically ill patients, treatments aimed at preventing acute kidney injury are warranted.

EA-230 is a novel pharmacological compound being developed for the treatment of systemic inflammatory states like sepsis, and for the treatment of inflammation associated organ dysfunction like acute kidney injury (AKI). It's a linear tetrapeptide derived from the human chorionic gonadotropin hormone (hCG). It has shown anti-inflammatory properties and protects against organ failure in several pre-clinical models of sepsis or systemic inflammation which will be described in more detail below. Most notably, EA-230 has shown marked protective effects in the kidney during abdominal sepsis in animals. As EA-230 attenuates the pro-inflammatory response in neutrophils and monocytes ex vivo, and neutrophil influx in tissues during systemic inflammation in vivo is abrogated, it is thought that EA-230 acts by protecting the host against the detrimental effects of neutrophils during acute systemic inflammatory diseases, thereby preventing organ damage, especially in the kidney.

Having performed extensive research into the pharmacology, pharmacokinetics and toxicology of EA-230, a first in human study was previously conducted with escalating single doses of EA-230, which showed that EA-230 was well tolerated up to i.v. doses of 30 mg/kg three times a day (daily dose of 90 mg/kg) for three days, and did not result in adverse events that were related to the study treatment. In a human model of systemic inflammation elicited by the administration of a low dose of endotoxin, EA-230 showed to attenuate the innate immune response at a single i.v. dose of 10 mg/kg, even though EA-230 was administered 30 minutes after endotoxin administration. A full dose- and concentration-response profile was not collected in that study. In addition, until now, only bolus administrations of EA-230 were tested, whereas in view of the short terminal half life of less than 15 minutes, a continuous administration of EA-230 over a longer time interval may be more effective.

For that reason, an additional phase I study in healthy volunteers is required to complete the profile of EA-230 response in inflammation before a dose or dose range can be chosen for a first 'prove-of-concept' study in patients. The safety profile of EA-230 has to be extended beyond the daily dose of 90 mg/kg addressed to date; the dose- and concentration response information collected during escalation will provide the dose for proof-of-concept testing in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 35 years inclusive
2. For part 2 only male
3. Subjects and their partners use a reliable way of contraception
4. BMI between 18 and 30 kg/m², with a lower limit of body weight of 50 kg
5. Healthy as determined by medical history, physical examination, vital signs, ECG, and clinical laboratory parameters

Exclusion Criteria:

1. Unwillingness to abstain from any medication, recreational drugs or anti-oxidant vitamin supplements during the course of the study and within 7 days prior to study Day 1.
2. Unwillingness to abstain from nicotine, or alcohol or within 1 day prior to study Day 1
3. Previous participation in a trial where LPS was administered
4. Surgery or trauma with significant blood loss or blood donation within 3 months prior to study Day 1
5. History, signs or symptoms of cardiovascular disease, in particular:

   * History of frequent vaso-vagal collapse or of orthostatic hypotension
   * Resting pulse rate ≤45 or ≥100 beats / min
   * Hypertension (RR systolic >160 or RR diastolic >90)
   * Hypotension (RR systolic <100 or RR diastolic <50)
   * conduction abnormalities on the ECG
6. Renal impairment: plasma creatinine >120 µmol/L
7. Liver function tests (alkaline phosphatase, AST, ALT and/or γ-GT) above 2x the upper limit of normal.
8. History of asthma
9. Atopic constitution
10. CRP above 2x the upper limit of normal, or clinically significant acute illness, including infections, within 2 weeks before administration of the study drug.
11. Treatment with investigational drugs or participation in any other clinical trial within 30 days prior to study drug administration.
12. Known or suspected of not being able to comply with the trial protocol.
13. Known hypersensitivity to any excipients of the drug formulations used.
14. Inability to personally provide written informed consent (e.g. for linguistic or mental reasons) and/or take part in the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability expressed in treatment related (serious) adverse events | total (S)AE's at day 14
  Adverse events include: clinically significant variation in vital signs compared to baseline (blood pressure and heart rate), local infusion reaction at site of i.v. IMP infusion, clinically significant changes in ECG compared to baseline and clinically significant deflections in laboratory parameters compared to baseline (Hb, Ht, Leucocytes, thrombocytes, Leucocyte differential blood count, sodium, potassium, creatinine, urea, alkaline phosphatase, ALT, AST, γGT, CK, CRP)

SECONDARY OUTCOMES:
Cytokines | at baseline (t=-1.5 and t=0), t=0.5, t=1, t=1,5 t=2, t=3, t=4, t=6, t=8 and t=24 hours after IMP and endotoxin administration
  Blood plasma levels of TNF-alfa, IL-6 and IL-10, IL-8, IL12-p70, IL-1RA, MCP-1, ICAM, VCAM, MIP1-alfa, MIP1-beta,
Pharmacokinetics - levels of EA-230 | at baseline, t=0.25, t=0.5, t=1, t=1,5 t=2, t=3, t=4, t=6, t=8 and t=24 hours after IMP and endotoxin administration
  Blood plasma levels of EA-230 and, if possible, metabolites
Pharmacokinetics - AUC | at baseline, t=0.25, t=0.5, t=1, t=1,5 t=2, t=3, t=4, t=6, t=8 and t=24 hours after IMP and endotoxin administration
  Area under the plasma concentration versus time curve (AUC) of EA-230 and, if possible, metabolites
Pharmacokinetics - peak plasma levels | at baseline, t=0.25, t=0.5, t=1, t=1,5 t=2, t=3, t=4, t=6, t=8 and t=24 hours after IMP and endotoxin administration
  Cmax of EA-230 and, if possible, metabolites
Pharmacokinetics - half life | at baseline, t=0.25, t=0.5, t=1, t=1,5 t=2, t=3, t=4, t=6, t=8 and t=24 hours after IMP and endotoxin administration
  plasma terminal t1/2 levels of EA-230 and, if possible, metabolites
Pharmacokinetics - distribution | at baseline, t=0.25, t=0.5, t=1, t=1,5 t=2, t=3, t=4, t=6, t=8 and t=24 hours after IMP and endotoxin administration
  Distibution volume (V) of EA-230 and, if possible, metabolites
Pharmacokinetics - Clearance | at baseline, t=0.25, t=0.5, t=1, t=1,5 t=2, t=3, t=4, t=6, t=8 and t=24 hours after IMP and endotoxin administration
  Clearance (Cl) of EA-230 and, if possible, metabolites
Renal function - GFR | one day before, during and one day after IMP en endotoxine administration
  GFR, measured by the clearance of iohexol, the endogenous creatinie clearance and estimated by the clearance of serum creatinine using MDRD.
Renal function - renal damage markers | at baseline(t=-1.5 and t=0), t=3, t=6, t=9, t=12 and t=24 hours after IMP en endotoxine administration
  Kidney injury markers measured by urine NGAL, KIM-1, L-FABP and plasma cystatin C.

CONTACTS AND LOCATIONS:
Overall Officials: P Pickkers, MD, Prof., Principal Investigator — Radboud University Medical Center
Locations (1):
- Intensive care, research unit, Radboud University Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] van Groenendael R, Kox M, Leijte G, Koeneman B, Gerretsen J, van Eijk L, Pickkers P. A randomized double-blind, placebo-controlled clinical phase IIa trial on safety, immunomodulatory effects and pharmacokinetics of EA-230 during experimental human endotoxaemia. Br J Clin Pharmacol. 2019 Jul;85(7):1559-1571. doi: 10.1111/bcp.13941. Epub 2019 May 23. PMID 30919998